CLINICAL TRIAL: NCT02929225
Title: Effect of Probiotics on Modulating the Bacterial Translocation and Improving Micro-inflammation in Hemodialysis Patients
Brief Title: Effectiveness of Probiotics to Treat End Stage Renal Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJTU1AF-CRS-2016-015
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Kidney Failure, Chronic
Keywords: bacterial translocation;micro-inflammation;hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifid Triple Viable Capsules (Experimental): BIFICO(Shanghai Sine Pharmaceutical Laboratories Co.Ltd,S10950032), A biological preparation composed of triple viable microbe(Live combined Bifidobacterium, Lactobacillus and enterococcus capsules)
  Interventions: Drug: Bifid Triple Viable Capsules
- placebo (Placebo Comparator): placebo is also manufactured by Sine Pharmaceutical Laboratories,but only contains starch.And placebo is the same as probiotics in appearance,odor,flavor and color.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Bifid Triple Viable Capsules — BIFICO is prescribed as a dose of 4 capsules twice daily in half hours after meals.
  Other Names: BIFICO,S10950032
  Arms: Bifid Triple Viable Capsules
Other: placebo — placebo is also prescribed as a dose of 4 capsules twice daily
  Other Names: placebo(Shanghai Sine Pharmaceutical Laboratories Co.Ltd)
  Arms: placebo

SUMMARY:
Intestinal microbiota has recently emerged as an important player in the progression and complications of chronic kidney disease(CKD). And drug therapy which selects the gut as a target has raised lots of concern. It has been reported that the composition of intestinal flora has changed in uremic patients. Specifically, imbalanced ecosystem has higher number of pathogens such as Clostridia, Enterobacteria,and lower number of beneficial microbes such as Lactobacilli and Bifidobacteria. This modification of intestinal flora can strongly increase transformation of amino acids into Uremic Retention solutes, e.g., indoxyl-sulfate (IS), p-cresyl sulfate (PCS), which are so called gut-derived uremic toxins. The dysbiosis also contributes to an increase in intestinal permeability by disrupting the colonic epithelial tight junction,which may subsequently lead to translocation of endotoxin and bacteria into the host's internal environment,resulting in systemic micro-inflammation.Also all of these can promote the progression of renal failure and the incidence of cardiovascular complications,renal osteodystrophy and anemia.Probiotics is defined by the World Health Organization as 'live microorganisms that, when administered in adequate amounts, confer a health benefit on the host'. Probiotics are being increasingly used for various pathologic conditions.It is said that probiotics have a therapeutic role in maintaining a metabolically balanced gastrointestinal tract (GIT).And in our previous study,the investigators found that in uremic rats,lactobacillus acidophilus can relieve bacterial translocation and decrease the level of inflammatory markers.So our study is mainly designed to investigate whether probiotics can modulate the balance of intestinal ecosystem, prevent the bacterial translocation from gut and alleviate the systemic inflammation in hemodialysis(HD) patients.

DETAILED DESCRIPTION:
This study is a single-centre, double-blind, placebo-controlled, randomised trial. Participants will undergo a 2 week run-in period, followed by randomisation to either probiotics supplements or placebo for 6 months. The study population are hemodialysis patients from Dialysis Department in First Affiliated Hospital of Xi'an Jiaotong University. The Dialysis Department have 400 patients who regularly come to receive dialysis therapy three times a week.It's relatively easy for us to follow up and collect data.Patients who meet the criteria and are able to provide informed consent will be recruited.Then computer-generated randomisation of participants to treatment order will be undertaken by an external statistical consultant. This process of allocation will conceal the randomisation order to researchers and participants. In addition, the supplements will be packed off-site with a generic label.

After randomization,baseline data will be collected and all participants will undergo face-to-face dietary education with a dietitian, incorporating standard hemodialysis education during the first week of run-in.In the week following, and throughout the intervention, patients will be encouraged to maintain stable protein and fibre intakes, with specific attention to maintaining the same sources of these nutrients.Participants' dietary intakes during the study will be assessed every month using a semi-quantitative food frequency questionnaire. And when the trial starts, questionnaires and biological samples will be performed and collected at the corresponding time. All serious adverse events will be reported to the ethics committee, whether deemed to be intervention related or not. Adherence to supplements will be measured by pill count every two weeks.

This study is an explorative clinical trial.And in the absence of any data about the effect of probiotics on hemodialysis patients intestinal and serum microbiota,sample size can't be calculated.Data will be reported as s mean±SD if normally distributed and as median(25-75% percentiles) if not. The Shapiro-Wilk test is performed to assess whether data are normally distributed. Statistical comparisons of normally distributed data are performed using Student's t-test. Mann-Whitney U-test is used to compare the rank variables measuring gastrointestinal symptoms in probiotics and placebo groups. The threshold for statistical significance is at p values <0.05. And an external statistical consultant from our Clinical Research Center will be involved in the data validation and analysis activities.

ELIGIBILITY:
Inclusion Criteria:

* maintenance hemodialysis patients(MHP),dialysis age>3 months;
* signed informed consent.

Exclusion Criteria:

* intolerance to whole milk and dairy products;
* patients with kidney transplant, with severe infections, sever heart disease and liver disease, malignancy, autoimmune disorders, severe malnutrition, or clinical conditions requiring artificial feeding;
* pregnant or nursing women;
* patients with known gastro-intestinal disease (i.e.,inflammatory bowel disease,crohn's disease,ulcerative colitis),receiving or have received radiation to the bowel or large bowel resection;
* use of antibiotics, prebiotics or probiotics in the past 4 weeks;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Gut microbiota | Change from Baseline in faeces bacterial genomic DNA at 6 months
  a faeces microbial analysis

SECONDARY OUTCOMES:
plasma detection of bacterial genomic DNA,plasma and fecal metabolomics | Change from Baseline in faeces bacterial genomic DNA at 6 months, fecal and plasma metabolomics at baseline and 6 months
plasma concentrations of inflammatory biomarkers(hs-C reactive protein,Interleukin(IL)-6,tumor necrosis factor(TNF)-α,endotoxin) | baseline,3 months and 6 months
Gastrointestinal Symptom Rating Scale (GSRS),SF-36 | baseline，3 and 6 months
  Monitor Gastrointestinal symptoms and life quality

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Jiang, professor, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The data including baseline characteristics of study population, blood biochemical index and main outcome measures may be made available.

REFERENCES:
- [Background] Hida M, Aiba Y, Sawamura S, Suzuki N, Satoh T, Koga Y. Inhibition of the accumulation of uremic toxins in the blood and their precursors in the feces after oral administration of Lebenin, a lactic acid bacteria preparation, to uremic patients undergoing hemodialysis. Nephron. 1996;74(2):349-55. doi: 10.1159/000189334. PMID 8893154
- [Background] Vaziri ND, Wong J, Pahl M, Piceno YM, Yuan J, DeSantis TZ, Ni Z, Nguyen TH, Andersen GL. Chronic kidney disease alters intestinal microbial flora. Kidney Int. 2013 Feb;83(2):308-15. doi: 10.1038/ki.2012.345. Epub 2012 Sep 19. PMID 22992469
- [Background] Koppe L, Mafra D, Fouque D. Probiotics and chronic kidney disease. Kidney Int. 2015 Nov;88(5):958-66. doi: 10.1038/ki.2015.255. Epub 2015 Sep 16. PMID 26376131
- [Background] Vaziri ND, Yuan J, Rahimi A, Ni Z, Said H, Subramanian VS. Disintegration of colonic epithelial tight junction in uremia: a likely cause of CKD-associated inflammation. Nephrol Dial Transplant. 2012 Jul;27(7):2686-93. doi: 10.1093/ndt/gfr624. Epub 2011 Nov 29. PMID 22131233
- [Background] Shi K, Wang F, Jiang H, Liu H, Wei M, Wang Z, Xie L. Gut bacterial translocation may aggravate microinflammation in hemodialysis patients. Dig Dis Sci. 2014 Sep;59(9):2109-17. doi: 10.1007/s10620-014-3202-7. Epub 2014 May 15. PMID 24828917
- [Background] Wang F, Jiang H, Shi K, Ren Y, Zhang P, Cheng S. Gut bacterial translocation is associated with microinflammation in end-stage renal disease patients. Nephrology (Carlton). 2012 Nov;17(8):733-8. doi: 10.1111/j.1440-1797.2012.01647.x. PMID 22817644
- [Background] Vanholder R, De Smet R, Glorieux G, Argiles A, Baurmeister U, Brunet P, Clark W, Cohen G, De Deyn PP, Deppisch R, Descamps-Latscha B, Henle T, Jorres A, Lemke HD, Massy ZA, Passlick-Deetjen J, Rodriguez M, Stegmayr B, Stenvinkel P, Tetta C, Wanner C, Zidek W; European Uremic Toxin Work Group (EUTox). Review on uremic toxins: classification, concentration, and interindividual variability. Kidney Int. 2003 May;63(5):1934-43. doi: 10.1046/j.1523-1755.2003.00924.x. PMID 12675874
- [Background] Dou L, Cerini C, Brunet P, Guilianelli C, Moal V, Grau G, De Smet R, Vanholder R, Sampol J, Berland Y. P-cresol, a uremic toxin, decreases endothelial cell response to inflammatory cytokines. Kidney Int. 2002 Dec;62(6):1999-2009. doi: 10.1046/j.1523-1755.2002.t01-1-00651.x. PMID 12427124
- [Background] Niwa T, Ise M, Miyazaki T. Progression of glomerular sclerosis in experimental uremic rats by administration of indole, a precursor of indoxyl sulfate. Am J Nephrol. 1994;14(3):207-12. doi: 10.1159/000168716. PMID 7977482
- [Background] Food and Agriculture Organsization. Guidelines for the Evaluation of Probiotics in Food. Joint FAO/WHO Working Group Report on Drafting Guidelines for the Evaluation of Probiotics in Food. Food and Agriculture Organization: London, 2002.
- [Background] Ebel B, Lemetais G, Beney L, Cachon R, Sokol H, Langella P, Gervais P. Impact of probiotics on risk factors for cardiovascular diseases. A review. Crit Rev Food Sci Nutr. 2014;54(2):175-89. doi: 10.1080/10408398.2011.579361. PMID 24188267
- [Background] Wei M, Wang Z, Liu H, Jiang H, Wang M, Liang S, Shi K, Feng J. Probiotic Bifidobacterium animalis subsp. lactis Bi-07 alleviates bacterial translocation and ameliorates microinflammation in experimental uraemia. Nephrology (Carlton). 2014 Aug;19(8):500-6. doi: 10.1111/nep.12272. PMID 24787732